CLINICAL TRIAL: NCT05978141
Title: The T-cell Lymphoma Master Repository (TCLMR): A Prospective Databank of Patients With T-cell Lymphoma With Clinical Annotation and Matched Tumor Specimens
Brief Title: A Registry for People With T-cell Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-190
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: T-cell Lymphoma; NK-Cell Lymphoma; T-cell Prolymphocytic Leukemia; T-cell Large Granular Lymphocytic Leukemia; Chronic Lymphoproliferative Disorder of NK Cells; Aggressive NK-cell Leukemia; Systemic Epstein-Barr Virus Positive T-Cell Lymphoproliferative Disease of Childhood (Disorder); Systemic Epstein Barr Virus Positive T-Cell Lymphoproliferative Disease of Childhood; Chronic Active EBV Infection of T-and NK-Cell Type, Systemic Form; Hydroa Vacciniforme-Like Lymphoproliferative Disorder; Adult T-cell Leukemia/Lymphoma; Extranodal NK/T-cell Lymphoma, Nasal Type; Enteropathy-associated T-cell Lymphoma; Monomorphic Epitheliotropic Intestinal T-Cell Lymphoma; Intestinal T-Cell Lymphoma, Not Otherwise Specified; Indolent T-Cell Lymphoproliferative Disorder of the Gastrointestinal Tract; Hepatosplenic T-cell Lymphoma; Subcutaneous Panniculitis-Like T-Cell Lymphoma; Mycosis Fungoides; Sezary Syndrome; Primary Cutaneous Anaplastic Large Cell Lymphoma; Primary Cutaneous T-cell Lymphoma; Primary Cutaneous CD8-Positive Aggressive Epidermotropic T-Cell Lymphoma; Primary Cutaneous Acral CD8-Positive T-Cell Lymphoma; Peripheral T-Cell Lymphoma, Not Otherwise Specified; Angioimmunoblastic T-cell Lymphoma; Follicular T-Cell Lymphoma; Nodal Peripheral T-Cell Lymphoma With TFH Phenotype; Anaplastic Large Cell Lymphoma, ALK-Positive; Anaplastic Large Cell Lymphoma, ALK-negative; Breast Implant-Associated Anaplastic Large Cell Lymphoma
Keywords: 23-190; T-cell lymphoma; Memorial Sloan Kettering Cancer Center; T-cell Lymphoma Master Repository; TCLMR
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, Prolymphocytic, T-Cell; Leukemia, Large Granular Lymphocytic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Enteropathy-Associated T-Cell Lymphoma; Subcutaneous panniculitis-like T-cell lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Primary Cutaneous Anaplastic Large Cell; Lymphoma, T-Cell, Cutaneous; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with T-Cell Lymphoma: Participants with pathologically-confirmed mature T- or natural killer (NK)-cell lymphoma
  Interventions: Other: Optional Blood Sample and Nail Sample

INTERVENTIONS:
Other: Optional Blood Sample and Nail Sample — Participants may provide optional research blood and nail samples for biobanking and future use

SUMMARY:
The purpose of this registry study is to create a database-a collection of information-for better understanding T-cell lymphoma. Researchers will use the information from this database to learn more about how to improve outcomes for people with T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adequate fresh or archival tumor biopsy or intent to obtain fresh tumor biopsy.
* Pathologically-confirmed mature T- or natural killer (NK)-cell lymphoma meeting one of the following diagnostic criterion (based on WHO classification and NCCN guidelines):

  * T-cell prolymphocytic leukemia
  * T-cell large granular lymphocytic leukemia
  * Chronic lymphoproliferative disorder of NK cells
  * Aggressive NK-cell leukemia
  * Systemic Epstein-Barr virus (EBV)-positive T-cell lymphoma of childhood
  * Chronic active EBV infection of T- and NK-cell type, systemic form
  * Hydroa vacciniforme-like lymphoproliferative disorder
  * Adult T-cell leukemia/lymphoma
  * Extranodal NK/T-cell lymphoma, nasal type
  * Enteropathy-associated T-cell lymphoma
  * Monomorphic epitheliotropic intestinal T-cell lymphoma
  * Intestinal T-cell lymphoma, not otherwise specified (NOS)
  * Indolent T-cell lymphoproliferative disorder of the gastrointestinal tract
  * Hepatosplenic T-cell lymphoma
  * Subcutaneous panniculitis-like T-cell lymphoma
  * Mycosis fungoides (limited to those with ≥ stage IB disease and those receiving active therapy)
  * Sézary syndrome
  * Primary cutaneous anaplastic large cell lymphoma (receiving systemic therapy)
  * Primary cutaneous Gamma-Delta T-cell lymphoma
  * Primary cutaneous CD8+ aggressive epidermotropic cytotoxic T-cell lymphoma
  * Primary cutaneous acral CD8+ T-cell lymphoma (receiving systemic therapy)
  * Peripheral T-cell lymphoma, not otherwise specified
  * Angioimmunoblastic T-cell lymphoma
  * Follicular T-cell lymphoma
  * Nodal peripheral T-cell lymphoma with TFH phenotype
  * Anaplastic large cell lymphoma, ALK-positive
  * Anaplastic large cell lymphoma, ALK-negative
  * Breast-implant associated anaplastic large cell lymphoma.
* NOTE: Patients with diagnoses of mycosis fungoides, primary cutaneous anaplastic large cell lymphoma, and/or primary cutaneous acral CD8+ T-cell lymphoma must be receiving systemic therapy.

Exclusion Criteria:

* Patients with of mycosis fungoides, primary cutaneous anaplastic large cell lymphoma, and/or primary cutaneous acral CD8+ T-cell lymphoma not receiving systemic therapy.
* Inability to collect prospective data, measure response, or perform adequate follow-up assessments in the clinical judgment of the treating physician. NOTE: Repository participation does not exclude participation in clinical trials, nor does existing clinical trial participation exclude enrollment in the study herein outlined.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants at Memorial Sloan Kettering Cancer Center (MSKCC) will be recruited through the Lymphoma service in the Department of Medicine and the Department of Pediatrics. Participants will be recruited at the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2030-07-27 (Estimated); Study Completion 2030-07-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants populating the T-cell Lymphoma Master Repository/TCLMR | 10 years
  To develop and populate a secure database comprised of patients with T-cell lymphomas with curated clinical characteristics and treatment outcomes matched to pathological biospecimens.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Horwitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (26):
- United States (26):
  - City of Hope Cancer Center (Data collection only), Duarte, California
  - UNIVERSITY OF CALIFORNIA SAN DIEGO (Data collection only), San Diego, California
  - University of California San Francisco (Data collection only), San Francisco, California
  - Stanford University Medical Center (Data collection only), Stanford, California
  - University of Colorado (Data Collection Only), Aurora, Colorado
  - Yale University (Data Collection Only), New Haven, Connecticut
  - University of Miami (Data Collection Only), Miami, Florida
  - Moffitt Cancer Center (Data Collection Only), Tampa, Florida
  - Emory University (Data Collection Only), Atlanta, Georgia
  - Northwestern Medicine (Data Collection), Chicago, Illinois
  - Massachusetts General Hospital (Data Collection Only), Boston, Massachusetts
  - Dana Farber Cancer Institute (Data Collection Only), Boston, Massachusetts
  - Mayo Clinic (Data Collection Only), Rochester, Minnesota
  - Washington University (Data Collection Only), St Louis, Missouri
  - University of Nebraska (Data collection only), Omaha, Nebraska
  - Memorial Sloan Kettering at Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Weill Cornell Medical Center (Data Collection Only), New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York
  - Ohio State University (Data Collection Only), Columbus, Ohio
  - University of Pennsylvania (Data Collection Only), Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital (Data collection only), Philadelphia, Pennsylvania
  - MD Anderson Cancer Center (Data Collection Only), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org